CLINICAL TRIAL: NCT04443439
Title: Head and Neck CTA Combined With Multimodal MRI to Assess the Risk of Cerebrovascular Disease
Brief Title: Assess the Risk of Cerebrovascular Disease
Status: Recruiting | Type: Observational
Sponsor: Tang-Du Hospital (Other)
Responsible Party: Principal Investigator, Wen Wang, MD & PhD, Director of radiology, Tang-Du Hospital
Other Study IDs: 2018LCYJ005
Record Dates: First submitted 2020-05-27; First posted 2020-06-23 (Actual); Last update posted 2022-10-25 (Actual); Status verified 2022-10

CONDITIONS: Cerebrovascular Disease
MeSH Terms: conditions — Cerebrovascular Disorders

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- No related neurological symptoms and transient ischemic attack: Mild stenosis group: CTA suggested carotid stenosis < 30%; Moderate stenosis group: CTA suggested carotid stenosis of 30-69%; Severe stenosis group: CTA indicated carotid stenosis ≥70%;
  Interventions: Device: GE Discovery MR750 3.0t superconducting MRI

INTERVENTIONS:
Device: GE Discovery MR750 3.0t superconducting MRI — T2WI, FLAIR, DWI, 3D BRAVO, 3D-ASL, rs-fMRI, DKI sequences to exclude other organic lesions

SUMMARY:
Intracranial artery stenosis is an important cause of ischemic stroke, but the degree of intracranial artery stenosis is not completely matched with the symptoms of ischemic stroke. Asymptomatic carotid stenosis (ACS) refers to does not appear related neurological symptoms of carotid stenosis and stroke or transient ischemic attack of carotid stenosis, did not happen cerebrovascular events such as stroke, but there have been a different degree of cognitive impairment, be badly in need of development of noninvasive imaging methods, objective evaluation of the ACS group cognitive impairment, and predict the ACS risk of ischemic stroke. Therefore, this topic proposed comprehensive cognitive assessment, CTA, double modal MRI techniques, clinical and biochemical indicator detection, mathematical modeling and statistical analysis techniques, assess the ACS group and normal person the cognitive ability, the difference of NVC and local perfusion, and follow-up ACS crowd of ischemic stroke and other cardiovascular events, discuss ACS and cognitive impairment, the correlation of NVC and local perfusion abnormalities, screening of radiographic predictor of ischemic stroke, and in the follow-up of ACS population in testing the sensitivity of the series of indicators and specific degrees.

ELIGIBILITY:
Inclusion Criteria:

1. Mild stenosis group: CTA suggested carotid stenosis < 30%;
2. Moderate stenosis group: CTA suggested carotid stenosis of 30-69%;
3. Severe stenosis group: CTA indicated carotid stenosis ≥70%;

Exclusion Criteria:

1. dementia, MMSE score < 21;
2. previous carotid stenosis related neurological symptoms or transient ischemic attack;
3. other craniocerebral lesions, such as craniocerebral trauma, tumor, inflammation, and complications of great vessels (cerebral infarction or cerebral malacia);
4. contraindications for MRI examination;
5. recent use of psychoactive drugs or hormones.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: No carotid stenosis - related neurological symptoms and transient ischemic attacks (50 patients in each group, 25 males and 25 females).
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2020-10-09 (Actual); Primary Completion 2026-11-15 (Estimated); Study Completion 2026-12-01 (Estimated)

PRIMARY OUTCOMES:
Dynamic change and correlation analysis of multi-dimensional features of ACS degree and cognitive impairment | 2020.01
  The Montreal cognitive assessment (MoCA) scale was used to evaluate the differences in cognitive function between ACS and the healthy control group in different dimensions, and the horizontal correlation analysis between ACS and cognitive impairment was conducted according to the dimensions of cognitive impairment and the degree of ACS.

CONTACTS AND LOCATIONS:
Locations (1):
- Wen Wang, Xi'an, China

DOCUMENTS (3):
  • Study Protocol: Study Protocol (2020-04-15): https://cdn.clinicaltrials.gov/large-docs/39/NCT04443439/Prot_000.pdf
  • Statistical Analysis Plan (2020-04-15): https://cdn.clinicaltrials.gov/large-docs/39/NCT04443439/SAP_001.pdf
  • Informed Consent Form (2020-04-15): https://cdn.clinicaltrials.gov/large-docs/39/NCT04443439/ICF_002.pdf